CLINICAL TRIAL: NCT06535854
Title: A Randomized Controlled Study of the Prevail Drug-Coated Balloon in Subjects With In-stent Restenosis and a Single Arm Prospectively Enrolled Study of the Prevail Drug-Coated Balloon for de Novo Lesions in Small Vessel Disease (Prevail Global).
Brief Title: Prevail Global Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDT22021
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease
Keywords: ISR; DNSV
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Masking only applies to the subjects in the ISR Cohort, subjects will be randomized at a 1:1 ratio to treatment with the Prevail DCB or the Agent DCB.
  Subjects in DNSV Cohort will be prospectively enrolled in the study and treated with Prevail DCB.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ISR Cohort Prevail DCB (Experimental): To evaluate the clinical safety and efficacy of the Prevail DCB in the treatment of ISR with coronary lesions previously treated with drug-eluting or bare metal stents in native coronary arteries.
  Interventions: Device: Prevail DCB; Device: Agent DCB
- DNSV Cohort (RVD 2.0 - 2.75mm) (Experimental): To evaluate the clinical safety and efficacy of the Prevail DCB as compared to a DES historical control in subjects undergoing PCI for de novo lesions in small vessel disease.
  Interventions: Device: Prevail DCB

INTERVENTIONS:
Device: Prevail DCB — The Prevail Paclitaxel-coated PTCA Balloon Catheter is intended for percutaneous transluminal coronary angioplasty (PTCA) in the coronary arteries with a vessel diameter from 2.00 mm to 4.00 mm to treat in-stent restenosis (ISR) and to treat de novo lesions in small vessel disease.
Device: Agent DCB — The Agent Paclitaxel-coated PTCA Balloon Catheter is intended for percutaneous transluminal coronary angioplasty (PTCA) in the coronary arteries with a vessel diameter from 2.00 mm to 4.00 mm to treat in-stent restenosis (ISR).
  Arms: ISR Cohort Prevail DCB

SUMMARY:
The purpose of the study is to evaluate the clinical safety and efficacy of the Prevail DCB.

DETAILED DESCRIPTION:
The Prevail Global study is a prospective, premarket, interventional, multi-center, global, dual cohort clinical study enrolling subjects undergoing percutaneous coronary intervention for in-stent restenosis (ISR Cohort) in a randomized controlled study of the Prevail Drug-Coated Balloon, and subjects undergoing percutaneous coronary intervention of the Prevail Drug-Coated Balloon for de novo lesions in small vessel disease (DNSV Cohort) in a single arm prospectively enrolled study.

In the ISR Cohort this will be accomplished by randomizing subjects to either a Prevail DCB arm or an Agent DCB arm to compare results of the treatment of ISR with coronary lesions previously treated with DES or BMS in native coronary arteries. In the DNSV Cohort this will be accomplished through collection of data to compare results of the Prevail DCB to a DES historical control in subjects undergoing PCI for de novo lesions in small vessel disease.

Subjects will be enrolled at approximately 65 study sites; the same study sites will be used for enrollment of both cohorts. The enrollment period is anticipated to be approximately 12 months. Subjects will remain in the study with follow-up clinical assessments through 5 years, study exit, or death, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Negative pregnancy test
* Stable or unstable angina, positive functional test, or stable NSTEMI
* Life expectancy >1 year
* Willing and able to cooperate with study procedures and required follow up evaluations

Exclusion Criteria:

* Known hypersensitivity or contraindication to antiplatelet medications or a sensitivity to contrast media which cannot be adequately pre-medicated
* History of an allergic reaction or significant sensitivity to paclitaxel or any other analogue or derivative
* Platelet count < 100,000 cells/mm³ or > 700,000 cells/mm³, or a white blood cell (WBC) count < 3,000 cells/mm³
* Renal insufficiency (or failure)
* Acute MI
* Previous PCI of the target vessel within 6 months prior to the procedure
* Planned PCI of any vessel within 30 days post-index procedure and/or planned PCI of the target vessel within 12 months post-procedure
* History of a stroke or transient ischemic attack (TIA)
* Active peptic ulcer or upper gastrointestinal (GI) bleeding
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Documented left ventricular ejection fraction (LVEF) <30%
* Planned surgery that would cause interruption in recommended DAPT duration per current guidelines
* Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints; or requires additional coronary angiography, IVUS or other coronary artery imaging procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1205 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
ISR Cohort Primary Analysis | 1 year post-procedure
  The TLF rate of the Prevail DCB arm at 12 months post procedure compared to the Agent DCB arm for non-inferiority
DNSV Cohort Primary Analysis | 1 year post-procedure
  The TLF rate of the Prevail DCB arm at 12 months post procedure compared to a DES historical control

SECONDARY OUTCOMES:
Acute success | hospital discharge, 30 days, and 6, 12, 24, 36, 48, and 60 months
  Acute success (device, lesion, and procedure) through hospital discharge only
All deaths | hospital discharge, 30 days, and 6, 12, 24, 36, 48, and 60 months
Cardiac death | hospital discharge, 30 days, and 6, 12, 24, 36, 48, and 60 months
All myocardial infarction (MI), including target vessel myocardial infarction (TVMI) | hospital discharge, 30 days, and 6, 12, 24, 36, 48, and 60 months
Clinically-driven target lesion revascularization (cd-TLR) defined as repeat PCI or CABG to the target lesion | hospital discharge, 30 days, and 6, 12, 24, 36, 48, and 60 months
Clinically-driven target vessel revascularization (cd-TVR) | hospital discharge, 30 days, and 6, 12, 24, 36, 48, and 60 months
Major adverse cardiac event (MACE) defined as composite of death, MI, or repeat cd-TLR | hospital discharge, 30 days, and 6, 12, 24, 36, 48, and 60 months
Target lesion failure (TLF) defined as composite of cardiac death, TVMI, or cd-TLR | hospital discharge, 30 days, and 6, 12, 24, 36, 48, and 60 months
Target vessel failure (TVF) defined as composite of cardiac death, TVMI, or cd-TVR | hospital discharge, 30 days, and 6, 12, 24, 36, 48, and 60 months
Target lesion thrombosis (TLT) (definite or probable) according to Academic Research Consortium (ARC) definition | hospital discharge, 30 days, and 6, 12, 24, 36, 48, and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, Principal Investigator — Piedmont Heart Institute; Bruno Scheller, Principal Investigator — University of Saarland; Azeem Latib, Principal Investigator — Montefiore Health System; Darren Mylotte, Principal Investigator — Galway University Hospitals
Locations (45):
- United States (45):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - Carondelet Saint Marys, Tucson, Arizona
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - Stanford Hospital & Clinics, Stanford, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - BayCare Health System, Clearwater, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - University of Miami Hospital, Miami, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Parkview Health, Fort Wayne, Indiana
  - Kansas City Heart Rhythm Institute (Midwest Heart and Vascular Specialist), Overland Park, Kansas
  - Ascension Via Christi Saint Francis, Wichita, Kansas
  - Saint Elizabeth Healthcare, Edgewood, Kentucky
  - Corewell Health, Grand Rapids, Michigan
  - Saint Joseph Mercy Ann Arbor, Ypsilanti, Michigan
  - M Health Fairview Clinic, Edina, Minnesota
  - CentraCare Heart & Vascular Center MN - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Lukes Mid America Heart Institute, Kansas City, Missouri
  - Providence Saint Patrick Hospital, Missoula, Montana
  - Virtua Our Lady of Lourdes Hospital, Camden, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - Kaleida Health, Buffalo, New York
  - Cumc/Nyph, New York, New York
  - Montefiore Medical Center, New York, New York
  - Saint Francis Hospital (Roslyn NY), Roslyn, New York
  - The Moses H Cone Memorial Hospital, Greensboro, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - The Lindner Research Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - UPMC Pinnacle Harrisburg Campus, Harrisburg, Pennsylvania
  - Rhode Island Hospital and Health Services - Lifespan, Providence, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - HCA Houston Medical Center, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Gundersen Lutheran, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kandzari DE, Latib A, Mylotte D, Ali ZA, Zaman A, Brar S, Parke M, Scheller B. Rationale and design of the prevail global trial program evaluating the prevail drug-coated balloon in patients with in-stent restenosis and de novo small vessel disease. Am Heart J. 2025 May;283:26-36. doi: 10.1016/j.ahj.2025.01.010. Epub 2025 Jan 23. PMID 39863032